CLINICAL TRIAL: NCT01800370
Title: The Effect of Mixed Exercise and Metabolic Stress Upon Pituitary Secretion in Relationship to Age in Healthy Men: a Pilot Study
Brief Title: The Effect of Mixed Exercise and Metabolic Stress in Relationship to Age in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Johannes D. Veldhuis, PI, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 12-007753
Record Dates: First submitted 2013-02-15; First posted 2013-02-27 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Healthy; Male
MeSH Terms: interventions — Sodium Chloride; Exercise; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hyperglycemia (Experimental): Hyperglycemia (rest controlled) will be induced by i.v. injection of 25 mL of dextrose 50% over 3 minutes with the subject supine. Includes blood draws and fasting requirements.
  Interventions: Drug: Hyperglycemia; Procedure: Blood Draws; Other: Fasting procedure
- Saline (Placebo Comparator): Saline (rest controlled) will be induced by i.v. injection of 25 mL of saline over 3 minutes with the subject supine. Includes blood draws and fasting requirements.
  Interventions: Drug: Saline; Procedure: Blood Draws; Other: Fasting procedure
- Exercise (Experimental): Monitored exercise of 7-minute biking, 2-minute arm weights and a blood draw at the 10-minute time point will be repeated 3 times,which takes 30 minutes.
  Bilateral arm curls begin at 20 pounds and decrease by 5 pounds as needed to sustain 2 minutes of exercise at a rate of 1 complete curl every 2 seconds.
  Includes blood draws and fasting requirements.
  Interventions: Other: Exercise; Procedure: Blood Draws; Other: Fasting procedure

INTERVENTIONS:
Drug: Hyperglycemia — Hyperglycemia (rest controlled) will be induced by i.v. injection of 25 mL of dextrose 50% over 3 minutes with the subject supine.
  Arms: Hyperglycemia
Drug: Saline — Saline (rest controlled) will be induced by i.v. injection of 25 mL of saline over 3 minutes with the subject supine.
  Arms: Saline
Other: Exercise — Monitored exercise of 7-minute biking, 2-minute arm weights and a blood draw at the 10-minute time point will be repeated 3 times,which takes 30 minutes.
  Bilateral arm curls begin at 20 pounds and decrease by 5 pounds as needed to sustain 2 minutes of exercise at a rate of 1 complete curl every 2 seconds.
  Arms: Exercise
Procedure: Blood Draws — Blood will be sampled every 10 min from 0700 to 1300 h. Each intervention will begin at 0800 h after 1 h of baseline sampling, and be completed by 0900 h. Intervention is followed by 4 additional h of sampling to capture recovery (total sampling 6 h). Ten-min samples are for Te, LH, ACTH, cortisol, and GH. Glucose will be checked every 30 min. At 07000 h an archival serum sample will be obtained for safety-monitoring purposes.
Other: Fasting procedure — Beginning at 1900 h on the evening prior to each study visit, subjects will remain fasting except for water, diet soda, and other non-caloric and non-caffeinated fluids, until 1300 h the next day.

SUMMARY:
Aging in men reduces the amount of luteinizing hormone (LH) and testosterone (Te) secreted in each burst. Stress-associated mechanisms introduced by acute illness and chronic disease decrease LH and Te secretion further. A major unresolved issue is whether the aging process heightens the negative effects of a stressor (whether physical or metabolic) upon LH and Te secretion. This study will assess LH and Te secretion in response to a physical stressor (maximal exercise) and a common metabolic stressor (hyperglycemia) as a function of age in healthy men ages 18-80 yr.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling, healthy men age 18 to 80
* Body-Mass Index (BMI) 18-30 kg/m2
* Willingness to provide written informed consent
* Physician acceptable screening ECG for participants 60 years and older

Exclusion Criteria:

* recent use of psychotropic or neuroactive drugs (within five biological half-live)
* obesity (outside weight range above)
* acute weight change (loss or gain of >2 kg in 6 weeks
* Laboratory test results not deemed physician acceptable
* triglycerides > 300
* BUN >30
* creatinine > 1.5 mg/dL
* liver functions tests twice upper limit of normal
* electrolyte abnormality
* anemia; hemoglobin < 12.0 gm/dL
* drug or alcohol abuse
* psychosis, depression, mania or severe anxiety
* acute or chronic organ-system disease
* endocrinopathy, other than primary thyroidal failure receiving replacement
* untreated osteoporosis
* nightshift work or recent transmeridian travel (exceeding 3 time zones within 7 days of admission)
* PSA > 4.0 ng/mL, History or suspicion of prostatic disease (elevated PSA,indeterminate nodule or mass, obstructive uropathy)
* History of carcinoma (excluding localized basal cell carcinoma removed or surgically treated with no recurrence
* History of thrombotic arterial disease (stroke, TIA, MI, angina) or deep vein thrombophlebitis
* History of CHF, cardiac arrhythmias, congential QT prolongation, and medications used to treat cardiac arrhythmias
* Gynecomastia > 2 cm, untreated
* Untreated gallbladder disease
* History of smoking greater than one ppd.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in Testosterone concentration after 30 minutes of exercise | 30 minutes after initiating exercise
  During the exercise visit subjects will perform an exercise test on a bike and lift weights with both arms for a total of 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Veldhuis, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States